CLINICAL TRIAL: NCT02620111
Title: Effect of Protein High in Leucine on Muscle Protein Balance in Elderly Patients: Acute Study With Protein-tracer-techniques
Brief Title: Protein Balance in Protein Supplemented Elderly Patients: Acute Study With Protein-tracer-techniques
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in recruiting frail subjects.
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Council for Strategic Research (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 44853
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2015-06

CONDITIONS: Elderly

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whey protein high leucine (Experimental): Subjects are supplemented water in a fasted state for 180 minutes while the isotopic tracer 15Nphenylalanin is infused. Subjects are supplemented with whey protein high in leucine from 180 - 360 minutes while the isotopic tracer 15Nphenylalanin is infused.
  Interventions: Dietary Supplement: Whey protein high in leucin
- Whey protein normal leucine (Active Comparator): Subjects are supplemented water in a fasted state for 180 minutes while the isotopic tracer 15Nphenylalanin is infused. Subjects are supplemented with whey protein normal in leucine from 180 - 360 minutes while the isotopic tracer 15Nphenylalanin is infused.
  Interventions: Dietary Supplement: Whey protein normal in leucin

INTERVENTIONS:
Dietary Supplement: Whey protein high in leucin — This Group is analysed for muscle protein synthesis and breakdown, mTor pathway signaling and Amino acid metabolism while supplemented first water then whey protein high in leucin
  Arms: Whey protein high leucine
Dietary Supplement: Whey protein normal in leucin — This Group is analysed for muscle protein synthesis and breakdown, mTor pathway signaling and Amino acid metabolism while supplemented first water then whey protein normal in leucin.
  Arms: Whey protein normal leucine

SUMMARY:
The aim of this study is to investigate potential protein synthesis effects of whey protein high in leucine compared to whey protein with normal leucin content in elderly patients in a acute crossover setting. We will use the method of a 2 X 3 h tracer infusing protocol with 15Nphenylalanine along with blood samples and muscle biopsies.

DETAILED DESCRIPTION:
Background: Improved muscle function/strength will enhance the quality of life of the more frail elderly population. Dietary proteins and amino acids act as anabolic substrates in muscles in elderly people. In particular the amino acid leucine is suggested to have an impact on muscle protein synthesis. In collaboration with the Danish dairy company Arla Foods we will use their conventional Whey protein and leucine enriched Whey protein in an acute study on elderly patients.

Our aim is to examine the acute effects of supplementation with whey protein high in leucine compared to whey protein with normal leucine content on muscle protein synthesis and protein balance in elderly patients.

Methods: We include 10 elderly patients, age 60-85 years in a randomized crossover study. The subjects will be recruited from the Osteoporosis Section at the Department of Endocrinology at Aarhus University Hospital. The subjects are their own controls in 2 x 1 day interventions A: whey protein high in leucine and B: whey protein with normal leucine content. Interventions are conducted with a 4 week washout period between them. On the intervention day postprandial protein synthesis rate will be measured over 2 X 3h using a tracer infusing protocol with 15Nphenylalanine along with blood samples and muscle biopsies. For analyzing steps of signaling in muscle protein synthesis initiated by leucine mammalian target of rapamycin (mTor) and sites downstream from mTor is quantified using western blotting. Whole body protein kinetics are calculated using the formula Q=i*Ei/Ep-i

ELIGIBILITY:
Inclusion criteria:

- Healthy elder people

Exclusion criteria:

* Liver and kidney disease.
* Known diabetes or Hgb1c ≥6,5% (≥48mmol/l).
* Severe heart disease (NYHA-Class >2).
* Oral corticosteroid treatment within the last 3 month.
* participation in other intervention studies within the last 4 weeks.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Protein balance | Protein balance is measured in a triplet from 160-180 minutes into the protein supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Jesper L Mehlsen, Phd student, Principal Investigator — University of Aarhus
Locations (1):
- Department of endocrinology, Aarhus University hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No